CLINICAL TRIAL: NCT01508052
Title: The Effects of Sequential Compression Device on Body Temperature During Propofol Anaesthesia: A Comparison With Elastic Stockings
Brief Title: Sequential Compression Device on Body Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Jeong Kwak, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GIRBA2628
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Hypothermia
Keywords: core temperature; sequential compression device; total intravenous anesthesia
MeSH Terms: conditions — Hypothermia | interventions — Stockings, Compression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequential compression device (Active Comparator): Apply sequential compression device during the thyroidectomy
  Interventions: Device: elastic stockings
- elastic stockings (Experimental): Apply elastic stockings during the thyroidectomy
  Interventions: Device: sequential compression device

INTERVENTIONS:
Device: sequential compression device — applying sequential compression device during the surgery
  Other Names: SCD
  Arms: elastic stockings
Device: elastic stockings — applying elastic stockings during the surgery
  Other Names: ES
  Arms: sequential compression device

SUMMARY:
We hypothesized that sequential compression device (SCD) compression system might induce more decreases on core temperature by increasing lower extremity blood flow. And, this study investigated the effects of SCD compression system on body temperature in patients during total intravenous anesthesia (TIVA) with propofol and remifentanil.

DETAILED DESCRIPTION:
Anaesthesia was induced and maintained with propofol and remifentanil. During the surgery, temperature was measured and recorded using oesophageal temperature and the calf-minus-toe skin-surface temperature gradient, respectively.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* 20-65 year
* patient who undergoing elective thyroidectomy

Exclusion Criteria:

* coronary occlusive disease
* peripheral vascular disease
* BMI > 30 kg/m2
* abnormal thyroid function test
* laparoscopic assisted thyroidectomy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jeong Kwak, Study Director — Gachon University Gil Medical Center
Locations (2):
- South Korea (2):
  - HKwak, Incheon
  - Gachon University Gil Medical Center, Incheon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequential Compression Device | Elastic Stockings
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequential Compression Device | Elastic Stockings | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.3) | 48.2 (11.5) | 48 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Core Body Temperature
Description: Core temperature and arteriovenous shunt in the lower leg was measured using oesophageal temperature and the calf-minus-toe skin-surface temperature gradient.
Time Frame: from baseline record core temperature every 15 minutes up to operative end
Measure: Mean (Standard Deviation); unit: degree C
Arm/Group | Sequential Compression Device | Elastic Stockings
Number analyzed (Participants) | 20 | 20
degree C
  baseline value | 36.4 (0.42) | 36.3 (0.43)
  end of operation vallue | 35.7 (0.43) | 35.6 (0.41)

ADVERSE EVENTS:
Arm/Group | Sequential Compression Device | Elastic Stockings
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes